CLINICAL TRIAL: NCT00593788
Title: The Gaps-in-Noise Test: Gap Detection Thresholds in Normal-Hearing Young Adults
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Samelli, Alessandra Giannella, University of Sao Paulo
Other Study IDs: 113 / 02; 113/02 de 03/13/2002
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Auditory Perception; Psychoacoustics
Keywords: GIN test; gap detection; temporal resolution; auditory perception; psychoacoustics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Normal-hearing adults between 18 and 31 years of age.

SUMMARY:
The aim of this study was to establish parameters for the Gaps-in-Noise test in normal-hearing young adults. One hundred subjects (50 males and 50 females) received an audiological evaluation to rule out hearing loss and auditory processing disorder. The Gaps-in-Noise test was then conducted on all subjects. The mean gap detection threshold was 4.19 msec. A psychometric function by gap duration was constructed, revealing that the percentage of correct responses was less than or equal to 5% for a gap duration of 2 msec, 10-30% for a gap duration of 3 msec, 60-70% for a gap duration of 4 msec, and over 96% for gap durations of 5 msec or longer. The results suggest that the data obtained can be applied as reference values for future testing. In the subjects evaluated, the Gaps-in-Noise test proved to be consistent with low variability.

ELIGIBILITY:
Inclusion Criteria:

Subject inclusion criteria were:

* all of the subjects have to have auditory thresholds lower than 20 dB HL at all of the frequencies evaluated (octave frequencies between 0.25 to 8 kHz), bilaterally;
* type A tympanometric curves with presented ipsilateral and contralateral acoustic reflexes;
* 95% or higher correct responses for each ear in the dichotic digit test.

Subject inclusion criteria also included negative histories for audiologic, otologic, head trauma, and neurologic involvement.

Exclusion Criteria:

* Hearing loss;
* Auditory processing disorder;
* Histories of audiologic, otologic, head trauma, and neurologic involvement.

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal-hearing adults between 18 and 31 years of age were evaluated, including 50 males (mean age 24.72 years) and 50 females (mean age 23.77 years). The youngest male subject was 18 years old, and the youngest female subject was 18.16 years old. In contrast, the oldest male subject was 31.5 years old, and the oldest female subject was 31.83 years old. All of the participants in the study were students or employees of the University of Guarulhos.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
gap detection test | half hour

CONTACTS AND LOCATIONS:
Overall Officials: alessandra G. Samelli, Doctor, Principal Investigator — Guarulhos University
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil